CLINICAL TRIAL: NCT02666560
Title: Does Increasing Auditory Cueing Affect Gait Parameters in Children With Cerebral Palsy During a Functional Task?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Collaborators: Gateshead Health NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 141A22
Record Dates: First submitted 2016-01-07; First posted 2016-01-28 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-04

CONDITIONS: Cerebral Palsy; Children
Keywords: Auditory Cueing; Gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auditory cueing at self paced cadence (Active Comparator): Participants performed a functional task with auditory cueing set at self paced cadence.
  Interventions: Device: Auditory Cueing
- Cueing at 20% above self paced cadence (Experimental): Participants performed a functional task with auditory cueing set at 20% above self paced cadence whilst performing a functional task.
  Interventions: Device: Auditory Cueing

INTERVENTIONS:
Device: Auditory Cueing — Auditory cueing set at different frequency rates

SUMMARY:
To determine the clinical efficacy of auditory cueing using a cross over design to investigate whether increasing auditory cueing frequency by 20% above self paced cadence affects gait parameters in children with Cerebral Palsy when performing a functional task.

DETAILED DESCRIPTION:
Introduction: Cerebral Palsy is a non progressive disorder occurring in early brain development, resulting in inefficient ambulatory pattern. The use of sensory cues to facilitate loco-motor activity has been suggested as providing the necessary trigger to synchronise movement with greater beneficial outcomes observed at higher frequency intensities within the adult population. Thus auditory cueing could have the potential to alter gait parameters during a functional task.

Aim: To explore if increasing auditory cueing frequency (AC20) affects gait during a functional task compared to auditory cueing at self-paced cadence (ACSC).

Method: Nineteen children with CP levels 1 and 2 on the Gross Motor Function Classification Scale participated using paired analysis. Outcomes were compared to the mean values for temporal spatial gait data within the conditions using a cross over design. TS data was obtained by using the GAITRite® walkway system whilst walking holding a cup.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cerebral Palsy aged 5 to 11 years old who were scored as levels 1 to 2 on the Gross Motor Function Classification Scale.
* Cognitive status average or above on the Weschler Intelligence Scale for children.
* Able to hear without the use of a hearing aid.

Exclusion Criteria:

* Hearing impairment that results in the use of a hearing aid.
* Walking with assistance of a mobility aid.
* Cardiovascular problems or other associated health problems which limits the child waking multiple times over the GAITRite®.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Walk-ley, Principal Investigator — University College, London; Ann Lyons, PHD, Study Chair — Northumberia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum PL, Walter SD, Hanna SE, Palisano RJ, Russell DJ, Raina P, Wood E, Bartlett DJ, Galuppi BE. Prognosis for gross motor function in cerebral palsy: creation of motor development curves. JAMA. 2002 Sep 18;288(11):1357-63. doi: 10.1001/jama.288.11.1357. PMID 12234229
- [Background] Kwak, E. (2007) Effect of rhythmic auditory stimulation on controlling stepping cadence of individuals with mental retardation and cerebral palsy. International journal of special education, vol 27, no 3, pp. 1-8.
- [Background] Kim SJ, Kwak EE, Park ES, Lee DS, Kim KJ, Song JE, Cho SR. Changes in gait patterns with rhythmic auditory stimulation in adults with cerebral palsy. NeuroRehabilitation. 2011;29(3):233-41. doi: 10.3233/NRE-2011-0698. PMID 22142756

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at an NHS FoundationTrust between March to April 2015. Twenty-six children with Cerebral Palsy who were currently on the paediatric physiotherapy caseload met the inclusion criteria, so were invited to participate. A total of nineteen children chose to participate in this research project.
Groups:
- Cueing Self Paced Then Cueing 20% Above Self Paced Cadence: Participants performed a functional task with auditory cueing set at self paced cadence. Five days following participants performed a functional task with auditory cueing set at 20% above self paced cadence.
  Auditory Cueing: This was was delivered by a metronome, which was set at a beat frequency rate that matched the participant's baseline cadence or 20% above baseline cadence.
- Cueing at 20% Above Self Paced Cadence Then Self Based Cadence: Participants performed a functional task with auditory cueing set at 20% above self paced cadence. Five days following participants performed a functional task with auditory cueing set at self paced cadence.
  Auditory Cueing: This was delivered by a metronome, which was set at a beat frequency rate 20% above baseline cadence or that matched the participant's baseline cadence.
Period: Condition 1 (1 Day)
Arm/Group | Cueing Self Paced Then Cueing 20% Above Self Paced Cadence | Cueing at 20% Above Self Paced Cadence Then Self Based Cadence
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0
Period: Condition 2 (1 Day)
Arm/Group | Cueing Self Paced Then Cueing 20% Above Self Paced Cadence | Cueing at 20% Above Self Paced Cadence Then Self Based Cadence
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants performed a functional task with auditory cueing set at self paced cadence and 20% above self paced cadence.
  Auditory Cueing: This was delivered by a metronome producing a beat which was set at the participant's baseline cadence or 20% above baseline cadence.
  This was a crossover design where participants completed both arms in the trial.
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 104.3 (25.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Step Length as Measured by the Gaitrite Walk-way System.
Description: The Gaitrite is a portable gait analysis walk-way system that enables the temprospatial measures of gait to be recorded. The temprospatial measure of length was recorded in centimetres.
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- ACSC: Auditory cueing at self paced cadence
- AC20: Auditory cueing set at 20% above self paced cadence
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
cm | 51.32 (6.42) | 53.36 (8.07)

2. Secondary Outcome: Velocity as Measured by the Gaitrite Walk-way System.
Description: The Gaitrite is a portable gait analysis walk-way system that enables the temprospatial measures of gait to be recorded. The temprospatial measure of velocity was recorded in cm's per second.
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- AC20: Auditory cueing at 20% above self paced cadence
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
cm/s | 98.62 (16.29) | 101.77 (21.08)

3. Secondary Outcome: Step Time as Measured by the Gaitrite Walk-way System.
Description: The Gaitrite is a portable gait analysis walk-way system that enables the temprospatial measures of gait to be recorded. The temprospatial measure of step time was recorded in seconds.
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
seconds | 0.53 (0.09) | 0.52 (0.08)

4. Secondary Outcome: Cadence as Measured by the Gaitrite Walk-way System.
Description: The Gaitrite is a portable gait analysis walk-way system that enables the temprospatial measures of gait to be recorded. The temprospatial measure of cadence was recorded in steps per minute.
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: steps per minute
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
steps per minute | 115.27 (15.75) | 117.09 (15.97)

5. Secondary Outcome: Time Spent in Double Support as Measured by the Gaitrite Walk-way System.
Description: The Gaitrite is a portable gait analysis walk-way system that enables the temprospatial measures of gait to be recorded. This was record in percentage of time spent in double support (%).
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
percentage of time | 0.30 (0.91) | 0.29 (0.09)

6. Secondary Outcome: Time Spent in Single Support as Measured by the Gaitrite Walk-way System.
Description: as for outcome 5
Time Frame: Data was collected at a single time point for each condition. Conditions occurred within a two week time period.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | ACSC | AC20
Number analyzed (Participants) | 19 | 19
percentage of time | 0.38 (0.05) | 0.39 (0.05)

ADVERSE EVENTS:
Time Frame: Two months on completion of the study
Description: All the participants were followed up during the routine physiotherapy review appointments upon completion of the study. No adverse events were reported.
Arm/Group | Auditory Cueing at Self Paced Cadence | Cueing at 20% Above Self Paced Cadence
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No